CLINICAL TRIAL: NCT07186140
Title: A Prospective Cohort Study to Explore Clinical Features, Prognosis, and Therapeutic Strategies in Patients With Acute Respiratory Distress Syndrome
Brief Title: Clinical Features, Treatments, and Outcomes in Acute Respiratory Distress Syndrome (ARDS-CTO)
Acronym: ARDS-CTO
Status: Not yet recruiting | Type: Observational
Sponsor: Jee Hwan Ahn (Other)
Responsible Party: Sponsor-Investigator, Jee Hwan Ahn, Assistant Professor, University of Ulsan College of Medicine; Director, Medical ICU, Asan Medical Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: 2025-0891
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute respiratory distress syndrome (ARDS)

SUMMARY:
The goal of this observational prospective cohort study is to explore the clinical characteristics, treatment strategies, and outcomes of adult patients with acute respiratory distress syndrome (ARDS) admitted to the medical intensive care unit of Asan Medical Center. The main questions it aims to answer are:

* What are the clinical features, current practices, and prognosis of ARDS patients in Korea?
* How do different mechanical ventilation settings affect ARDS patient outcomes?

Participants will:

* Be screened at medical ICU admission for eligibility according to the Berlin definition of ARDS.
* Have demographic, clinical, laboratory, and ventilator data collected from bedside monitoring devices and electronic health records during their ICU stay.
* Complete a quality-of-life questionnaire (EQ-5D) at hospital discharge if they survive.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Receiving respiratory support with one of the following:
* High-flow nasal oxygen (HFNO) at a flow rate ≥ 30 L/min,
* Noninvasive ventilation (NIV) with positive end-expiratory pressure (PEEP) of ≥ 5 cm H₂O, or
* Invasive mechanical ventilation with PEEP of ≥ 5 cm H₂O.
* Within 48 hours before or after eligibility screening, the following criteria must be met:
* PaO₂/FiO₂ ≤ 300 mmHg under the above respiratory support.
* Bilateral opacities on chest radiograph or computed tomography, not fully explained by effusions, lobar/lung collapse (atelectasis), or pulmonary nodules/masses.
* Respiratory failure not fully explained by cardiac failure or fluid overload; when no clear ARDS risk factor is identified, an objective assessment (e.g., echocardiography) is required to exclude hydrostatic edema.

Exclusion Criteria:

* Refusal of informed consent by the patient or a legally authorized representative.
* Chronic respiratory failure, defined as:
* Patients receiving long-term oxygen therapy or home mechanical ventilation (except for CPAP used solely for obstructive sleep apnea), or
* Outpatients with PaCO₂ > 60 mmHg.
* Diffuse alveolar hemorrhage.
* Interstitial lung disease.
* Moribund patients expected to survive < 24 hours.
* Patients expected to require high-flow nasal oxygen or mechanical ventilation for < 48 hours.
* Patients with a decision to withhold life-sustaining treatment (except those for whom full support is provided other than cardiopulmonary resuscitation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants from among patients with acute respiratory failure who are admitted to the medical intensive care unit of Asan Medical Center in Seoul, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days within 28 days | From enrollment to Day 28
  Number of days alive and free from invasive mechanical ventilation during the first 28 days after enrollment. Patients who die within 28 days will be assigned zero ventilator-free days.

SECONDARY OUTCOMES:
28-day mortality | From enrollment to Day 28
  All-cause mortality within 28 days after enrollment.
90-day mortality | From enrollment to Day 90
  All-cause mortality within 90 days after enrollment.
ICU mortality | From enrollment until ICU discharge, up to 90 days
  Death occurring during the index ICU stay.
Hospital mortality | From enrollment until hospital discharge, up to 90 days
  Death occurring during the index hospital admission.
Duration of invasive mechanical ventilation | From enrollment to Day 90
  Total number of days patients require invasive mechanical ventilation.
ICU length of stay | From enrollment until ICU discharge, up to 90 days
  Total number of days spent in the ICU.
Hospital length of stay | From enrollment until hospital discharge, up to 90 days
  Total number of days spent in the hospital.
Ventilator-associated pneumonia (VAP) | From enrollment until ICU discharge, up to 90 days
  Incidence of VAP diagnosed according to standard clinical criteria during the index ICU stay.
Central line-associated bloodstream infection (CLABSI) | From enrollment until ICU discharge, up to 90 days
  Incidence of CLABSI diagnosed according to CDC/NHSN criteria during the index ICU stay.
Barotrauma | From enrollment until ICU discharge, up to 90 days
  Incidence of pneumothorax, pneumomediastinum, or subcutaneous emphysema documented by imaging or clinical assessment during the index ICU stay.
Quality of life at hospital discharge | From enrollment until hospital discharge, up to 90 days
  Health-related quality of life assessed using the 5-level European Quality of Life 5 Dimensions version (EQ-5D-5L) questionnaire at the time of hospital discharge for survivors. Scores range from -0.066 to 1.0 (based on Korean Time Trade-Off value set), with higher scores indicating better health status.
Disposition at hospital discharge | From enrollment until hospital discharge, up to 90 days
  Patient's destination at hospital discharge (e.g., home, rehabilitation, long-term care facility, or death).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided